CLINICAL TRIAL: NCT03868215
Title: Use of Plasma ctDNA Methylation Haplotypes in Detecting Local Residual or Lymph Node Metastasis: a Prospective, Clinical Study
Brief Title: Use of Plasma ctDNA Methylation Haplotypes in Detecting Local Residual or Lymph Node Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guoxiang Cai, Professor, Fudan University
Other Study IDs: FDLNM-CGX
Record Dates: First submitted 2018-11-09; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer; Lymph Node Metastases
Keywords: Colorectal Cancer; Lymph Node Metastases; Local Residual
MeSH Terms: conditions — Colorectal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with endoscopically removed malignant polyps: Patients with endoscopically removed malignant polyps
  Interventions: Diagnostic Test: Next-generation sequencing (NGS)

INTERVENTIONS:
Diagnostic Test: Next-generation sequencing (NGS) — NGS test for colorectal tumor-specific plasma ctDNA methylation markers prior to endoscopy and before surgical resection.

SUMMARY:
This is a prospective, clinical study. This study is to evaluate the sensitivity of plasma ctDNA methylation haplotypes in detecting local residual or lymph node metastasis.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer worldwide, the second deadliest cancer in the United States. DNA methylation is a commonly used biomarker for non-invasive CRC detection in plasma. The low sensitivity of blood-based tests is due to several limitations of detecting ctDNA in early-stage cancer. We developed and validated a high-throughput methylation-based blood test highly sensitive for colorectal cancer and precancerous lesions. This previously established colorectal tumor-specific plasma ctDNA methylation markers (diagnostic model established by next-generation sequencing of 2181 gene loci methylation) had a high sensitivity in CRC patients and a high specificity in healthy individuals in a large retrospective sample study. This prospective, clinical study is to further evaluate the sensitivity of plasma ctDNA methylation haplotypes in detecting local residual or lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endoscopically removed malignant polyps.
* Male or female ≥ 18 years of age on the day of signing informed consent.
* Patients who received surgical resection following removal of malignant polyps by colonoscopy.
* Patients must have a performance status of ≤1 on the ECOG Performance Scale.
* Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study

Exclusion Criteria:

* Patients received adjuvant treatment prior to the surgical resection.
* Patients received blood transfusion two weeks before or during the surgical resection.
* Patients with unresected advanced colorectal adenoma.
* Patients who are positive for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C.
* Patients who are pregnant.
* Patients who are alcoholic or drug abusers.
* Patients with a history or current evidence of any condition or abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endoscopically removed malignant polyps must have baseline evaluations performed prior to the study and must meet all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 2 years
  The sensitivity of plasma ctDNA methylation haplotypes in detecting local residual or lymph node metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China